CLINICAL TRIAL: NCT01598818
Title: First-Sight Refractive Error Correction in the Developing World
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0553-11-FB
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Vision Loss
Keywords: Vision Nearsighted; Vision Farsighted
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Visual acuity: Comparison of best visual acuity and refraction using the First Sight Refractive System with autorefraction in subjects with refractive error.

SUMMARY:
The aim of this study is to test the efficacy of the First-Sight refractive kit designed to provide refractive correction of simple hyperopia, myopia and astigmatism with autorefraction.

DETAILED DESCRIPTION:
In remote and underserved areas, a patient may have limited or no access to eye specialists or healthcare facilities that offer equipment to provide standard refraction and purchase corrective lenses. First Sight Refracting system (FSR) is designed specifically to be used in remote and underserved areas. FSR is not considered the standard of care in the US. FSR is a portable refraction and lens-frame dispensing system with low cost of production. As a kit, it contains +/- 6.00 diopters of corrective lenses, color coordinated flipper, - 1.25 diopter astigmatism lens, visual acuity chart, astigmatic eye chart, measuring tape to measure the distance of the subject to the eye charts, pupillary distance ruler to measure for the frame size of the glasses to be dispensed, and lint free gloves. The kit comes with two standard frames. The corrective lenses are designed to be placed in the frames that can be readily dispensed to the patient after the refraction is done. The refraction technique is simple and straightforward and any healthcare worker in remote and underserved areas can provide the test and dispense glasses at no cost.

This is the third phase of First Sight refractive study to be done in Haiti. Adult and children subjects will be recruited during their routine examinations and/or visual acuity screenings at the Justinien Hospital. The proposed study will compare the visual acuity measurements obtained from the First Sight refraction system (test procedure) with the visual acuity measurements obtained from the autorefraction (standard care). The international study will recruit 150 subjects which will test FSR's effectiveness as a refracting tool of choice to be used in remote and underserved areas. Data from this study will be compared with the US studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 7 years of age and older
* Healthy subjects with no known ocular trauma, no surgery, ocular disease or pathology that would prevent obtainment of best correctable visual acuity to 20/30.

Exclusion Criteria:

* Refractive error greater than (+)/(-) 6.00 diopter, or astigmatism greater than 1.50 diopters.
* Known ocular (corneal, lenticular, vitreal, or retinal) pathology that may limit best correctable visual acuity.

Ages: 7 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Population with refractive error between -4.50 to +4.50 diopter spherical error and astigmatism up to 1.50 diopters.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-05-11 (Actual); Primary Completion 2014-01-13 (Actual); Study Completion 2014-01-13 (Actual)

PRIMARY OUTCOMES:
To compare the best visual acuity and refraction results using the First Sight Refraction System to standard auto-refraction in subjects with hyperopia. | 1 month
  A refractive error of +0.50 to +4.50 diopter spherical error and asitgmatism of 1.50 diopters will be assessed.

SECONDARY OUTCOMES:
To compare the best visual acuity and refraction results using the First Sight Refractive System to autorefraction in myopia. | 1 month
  A refractive error of -0.50 to -4.50 diopter spherical error and up to 1.50 astigmatism will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Feilmeier, MD, Principal Investigator — University of Nebraska Medical Center, Department of Ophthalmology and Visual Sciences
Locations (2):
- University of Nebraska Medical Center, Department of Ophthalmology, Omaha, Nebraska, United States
- Justinien Hospital, Cap-Haïtien, Haiti